CLINICAL TRIAL: NCT02744768
Title: D-ALBA Front-Line Sequential Treatment of Adult Philadelphia Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia (ALL) Patients With Dasatinib and the Bispecific Monoclonal Antibody Blinatumomab
Brief Title: D-ALBA Frontline Sequential Dasatinib and Blinatumomab in Adult Philadelphia Positive Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL2116
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia, adult, dasatinib, blinatumomab
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib; blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Adult Ph+ ALL (≥18 years old, with no upper age limit) patients will begin treatment with Dasatinib, 140 mg/day, from day 1 to day +84. Prednisone (PDN) will be administered from day -6 to day +0 (during which the presence of the BCR/ABL1 alteration will be established), at escalating doses up to 60 mg/m2; PDN will be continued up to day +24 and progressively tapered up to day +31.
  HLA typing will be performed immediately after the diagnosis for eligible patients.
  MRD will be evaluated by RT-PCR at fixed time points (days +22, +45, +57) during the induction and at day +85, the latter for molecular response evaluation.
  Interventions: Drug: Dasatinib; Drug: Blinatumomab

INTERVENTIONS:
Drug: Dasatinib — Adult Ph+ ALL (≥18 years old, with no upper age limit) patients will begin treatment with Dasatinib, 140 mg/day, from day 1 to day +84.
Drug: Blinatumomab — Upon induction:
  patients in CHR will receive Blinatumomab at a dose of 15 µg/m²/day as continuous intravenous infusion (CIVI) at a constant flow rate for four weeks, followed by a two-week infusion-free interval, defined as one treatment cycle. At least 2 cycles should be administered, up to a maximum of 5 cycles, if deemed necessary.

SUMMARY:
This study aims at exploring the activity of a frontline approach based on dasatinib plus steroids administration as induction treatment, followed by the infusion of Blinatumomab, in adult Ph+ ALL.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed adult B-precursor Ph+ ALL patients.
* Age greater or equal to18 years,
* Signed written informed consent according to ICH/EU/GCP and national local laws.
* ECOG Performance Status 0 or 1 and/or WHO performance status less or equal to 2.
* Renal and hepatic function as defined below:

  * AST (GOT), ALT (GPT), and AP <2 x upper limit of normal (ULN).
  * Total bilirubin <1.5 x ULN.
  * Creatinine clearance equal or greater than 50 mL/min.
* Pancreatic function as defined below:

  * Serum amylase less or equal to 1.5 x ULN
  * Serum lipase less or equal to1.5 x ULN.
* Normal cardiac function.
* Negative HIV test, negative HBV DNA and HCV RNA.
* Negative pregnancy test in women of childbearing potential.
* Bone marrow specimen from primary diagnosis available.

Exclusion Criteria:

* History of or current relevant CNS pathology (current ≥grade 2 epilepsy, seizure, paresis, aphasia, clinically relevant apoplexia, severe brain injuries, dementia, Parkinson's disease, organic brain syndrome, psychosis).
* Impaired cardiac function, including any one of the following:

  * LVEF <45% as determined by MUGA scan or echocardiogram.
  * Complete left bundle branch block.
  * Use of a cardiac pacemaker.
  * ST depression of >1mm in 2 or more leads and/or T wave inversions in 2 or more contiguous leads.
  * Congenital long QT syndrome.
  * History of or presence of significant ventricular or atrial arrhythmia.
  * Clinically significant resting bradycardia (<50 beats per minute).
  * QTc >450 msec on screening ECG (using the QTcF formula).
  * Right bundle branch block plus left anterior hemiblock, bifascicular block.
  * Myocardial infarction within 3 months prior to starting Dasatinib.
  * Angina pectoris.
* Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Dasatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* History of or current autoimmune disease.
* Systemic cancer chemotherapy within 2 weeks prior to study.
* Known hypersensitivity to immunoglobulins or to any other component of the study drug formulation.
* Active malignancy other than ALL with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix.
* Active infection, any other concurrent disease or medical conditions that are deemed to interfere with the conduct of the study as judged by the investigator.
* Nursing women or women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least 3 months thereafter or male patients not willing to ensure effective contraception during participation in the study and at least three months thereafter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who achieve Minimal Residual Disease (MRD) negativity upon treatment | After 11 months from study entry
  In particular, after 2 cycles of blinatumomab. Minimal Residual Disease (MRD) negativity is intended as Complete Molecular Remission (CMR)

SECONDARY OUTCOMES:
Number of patients completing the 2 cycles of blinatumomab and alive in first complete hematologic remission (CHR) | From day +85 at 12 months
Number of patients at Complete Molecular Response (CMR) | At day +22, +45, +57 and +85 from study entry
Number of months of the CMR | At 12 and 24 months
Number of patients in Overall Survival (OS) | At 12 and 24 months
Number of grade >3 adverse events | At 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foà, Study Chair — Policlinico Umberto I, Hematology Department.
Locations (34):
- Italy (34):
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - Az.Ospedaliera S.G.Moscati, Avellino
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Azienda Ospedaliera - Papa Giovanni XXIII, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Unità di Ricerca e di Malattie del sangue - Ematologia San Luca Vecchio Pad. 16 - 1° Piano, Florence
  - Unità Operative Complesse di Ematologia 1 e 2 Centro Trapianti di Midollo dell'IRCCS AOU San Martino-IST, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - U.O. di Ematologia- Ospedale dell'Angelo - Mestre, Mestre
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Ospedale Niguarda " Ca Granda" - SC Ematologia Blocco SUD, Ponti Est, Scala E, 4° piano, Milan
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - U.O. di Oncoematologia -plesso ospedaliero "A. Tortora" di Pagani, Pagani
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - UOC Medicina Trasfusionale e Cellule Staminali Azienda Ospedaliera San Camillo Forlanini, Roma
  - Policlinico Umberto I, Hematology Department, Rome
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Rome
  - Sezione di Ematologia Cancer Center Humanitas, Rozzano
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Struttura Complessa a Dir. Universitaria-Ematologia e Terapie Cellulari- A.S.O. Ordine Mauriziano, P.O. Umberto I-Ospedale Torino, Torino
  - Struttura Complessa a Dir. Universitaria-Ematologia e Terapie Cellulari- A.S.O. Ordine Mauriziano, P.O. Umberto I-Ospedale, Torino
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foa R, Bassan R, Elia L, Piciocchi A, Soddu S, Messina M, Ferrara F, Lunghi M, Mule A, Bonifacio M, Fracchiolla N, Salutari P, Fazi P, Guarini A, Rambaldi A, Chiaretti S. Long-Term Results of the Dasatinib-Blinatumomab Protocol for Adult Philadelphia-Positive ALL. J Clin Oncol. 2024 Mar 10;42(8):881-885. doi: 10.1200/JCO.23.01075. Epub 2023 Dec 21. PMID 38127722
- [Derived] Foa R, Bassan R, Vitale A, Elia L, Piciocchi A, Puzzolo MC, Canichella M, Viero P, Ferrara F, Lunghi M, Fabbiano F, Bonifacio M, Fracchiolla N, Di Bartolomeo P, Mancino A, De Propris MS, Vignetti M, Guarini A, Rambaldi A, Chiaretti S; GIMEMA Investigators. Dasatinib-Blinatumomab for Ph-Positive Acute Lymphoblastic Leukemia in Adults. N Engl J Med. 2020 Oct 22;383(17):1613-1623. doi: 10.1056/NEJMoa2016272. PMID 33085860
- See also: GIMEMA Foundation website — http://www.gimema.it

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT02744768/SAP_000.pdf
  • Study Protocol (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT02744768/Prot_001.pdf